CLINICAL TRIAL: NCT05834933
Title: Effects of Risk Assessment and Counselling on Adherence to Risk Reduction Recommendations Among Female Relatives of Breast Cancer Patients in Southwestern Nigeria
Brief Title: Nigerian Breast Cancer Risk-Reduction Study
Acronym: NBCRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ibadan (Other)
Collaborators: Lagos State University Teaching Hospital (LASUTH) (Unknown); Obafemi Awolowo University Teaching Hospital (Other); Lagos University Teaching Hospital (LUTH) (Unknown); University College Hospital, Ibadan (Other)
Responsible Party: Principal Investigator, Agwai Celia Imaria, Epidemiologist, University of Ibadan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: NHREC/05/01/2008a
Record Dates: First submitted 2023-03-05; First posted 2023-04-28 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Risk Reduction Behavior; Breast Cancer; Health Behavior; Health Care Utilization; Health Knowledge, Attitudes, Practice
Keywords: Breast cancer; First-degree relatives; Breast cancer prevention; Risk assessment; Risk counselling; Southwest Nigeria
MeSH Terms: conditions — Risk Reduction Behavior; Breast Neoplasms; Health Behavior; Patient Acceptance of Health Care; Behavior | interventions — Risk Assessment; Counseling

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants, Data collectors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (SC) (No Intervention): Participants received one-on-one breast cancer awareness education; one-on-one monthly Breast Self-Examination (BSE) training; general breast cancer screening recommendations; and general lifestyle modification recommendations
- SC + Risk assessment and counselling (Experimental): Participants received Standard care as described in the SC arm above in addition to individualized breast cancer risk assessment, individualized breast cancer risk counseling, and lifestyle risk reduction recommendations
  Interventions: Behavioral: Individualized breast cancer risk assessment; Behavioral: Individualized breast cancer risk counselling

INTERVENTIONS:
Behavioral: Individualized breast cancer risk assessment — Individualized breast cancer risk assessment: The Nigerian Breast Cancer Study (NBCS) absolute risk prediction model was used to predict the 5-year and lifetime breast cancer risks of the participants. The model utilized individual breast cancer risk factors.
  Other Names: Risk assessment
  Arms: SC + Risk assessment and counselling
Behavioral: Individualized breast cancer risk counselling — Individualized breast cancer risk counselling: The Principal Investigator (PI) and other trained risk counsellors discussed the results of the NBCS risk prediction model with participants and counselled them about the risk of developing breast cancer. The
  Other Names: Counseling
  Arms: SC + Risk assessment and counselling

SUMMARY:
The study will be a randomized controlled trial. The aim of the study is to determine the Breast Cancer (BC) risk and to evaluate the effect of BC risk counseling on lifestyle changes and adherence to risk-reduction practices among first-degree female relatives of BC patients in South-West Nigeria. This study's research questions are:

* What are the Nigeria Breast Cancer Study (NBCS) and Gail models estimates of the BC risk of first-degree female relatives of BC patients in South-West, Nigeria?
* What are the effects of BC risk assessment and counseling on adherence to breast screening recommendations among first-degree female relatives of BC patients in South-West, Nigeria?
* What are the effects of BC risk assessment and counseling on adherence to lifestyle risk reduction recommendations among first-degree female relatives of BC patients in South-West, Nigeria?
* What is the knowledge, attitudes, and perception of first-degree female relatives of BC patients in South-West Nigeria towards genetic testing and BC etiology?
* What factors predict breast screening among first-degree female relatives of BC patients in South-West Nigeria?
* What factors predict the time to first BC screening (post-intervention) among first-degree female relatives of BC patients in South-West Nigeria?

Participants will be randomized into the control arm (standard care) and intervention arms of the study. The intervention arm of the study will have a BC risk assessment followed by individualized BC risk counseling. In addition, the intervention arm will receive BC awareness and MammaCare® BSE training. The control arm will receive only standard care comprising BC awareness and MammaCare® BSE training. Both study arms will receive BC screening recommendations and lifestyle modification recommendations.

We hope that the BC risk counseling will improve BC screening practices and modification of risk behaviors and this hypothesis will be tested.

ELIGIBILITY:
Inclusion Criteria:

1. First-degree female relatives of histologically diagnosed BC patients in the study sites
2. Women aged 20 to 75 years of age
3. Willingness to be contacted after six months for follow-up

Exclusion Criteria:

1. Personal history of BC
2. Previous exposure to breast cancer risk assessment and counselling
3. Absence of intact breasts

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — For this study, first-degree female relatives are mothers, sisters, and daughters of BC patients
Enrollment: 719 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Effects of BC risk assessment and counselling on adherence to breast screening recommendations among first-degree female relatives of BC patients in South-West Nigeria | 6 months
  Questionnaire will be administered to the participants to determine the effects of the intervention on adherence to breast screening practices
Effects of BC risk assessment and counselling on adherence to lifestyle risk reduction recommendations among first-degree female relatives of BC patients in South-West, Nigeria | 6 months
  Questionnaire will be administered to the participants to determine the effects of the intervention on adherence to lifestyle risk reduction practices
Predictors of BSE among first-degree female relatives of BC patients in South-West Nigeria | 6 months
  Statistical analysis will be carried out to determined the independent variables predicting BSE
Predictors of time to first BC screening post-intervention among first-degree female relatives of BC patients in South-West Nigeria | Baseline
  Statistical analysis will be carried out to determined the independent variables predicting first time to BC screening

SECONDARY OUTCOMES:
Determine the perception of familial BC risk among first-degree female relatives of BC patients in South-West Nigeria. | Baseline
  Semi-structured questionnaires will be used to determine the perception of familial BC risk among participants
Determine the knowledge of familiar BC risk among first-degree female relatives of BC patients in South-West Nigeria. | Baseline
  Semi-structured questionnaires will be used to determine the knowledge of familiar BC risk among participants
Determine the knowledge, attitude, and perception towards genetic testing and BC aetiology among first-degree female relatives of BC patients in South-West Nigeria | Baseline
  Semi-structured questionnaires will be used to determine the knowledge, attitude, and perception towards genetic testing and BC aetiology among participants

CONTACTS AND LOCATIONS:
Overall Officials: OLADOSUN A OJENGBEDE, FMCOG, FWACS, FICS, M.B.B.S, Principal Investigator — CENTER FOR POPULATION AND REPRODUCTIVE HEALTH (CPRH), UNIVERSITY COLLEGE HOSPITAL, IBADAN; OLADELE O.O KALE, B.A, M.B, B.Ch, B.A.O, Principal Investigator — University of Ibadan; IKEOLUWAPO O. AJAYI, MBBS; PhD, Principal Investigator — University of Ibadan; CELIA IMARIA AGWAI, M.P.H; Ph.D., Principal Investigator — University of Ibadan; DEZHENG HUO, PhD, Study Director — University of Chicago; OLUFUNMILAYO OLOPADE, M.D., F.A.C.P, Study Chair — University of Chicago
Locations (4):
- Nigeria (4):
  - Obafemi Awolowo University Teaching Hospital Complex (OAUTHC), Ile-Ife, Osun State
  - University College Hospital (UCH), Ibadan, Oyo State
  - Lagos State University Teaching Hospital (LASUTH), Lagos
  - Lagos University Teaching Hospital (LUTH), Lagos

IPD SHARING:
Plan to Share IPD: No